CLINICAL TRIAL: NCT02803619
Title: A Multi-center Prospective Observational Biomarker Study on EGFRm+ Non-small Cell Lung Cancer Patients With Leptomeningeal Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wang mengzhao, Professor, Peking Union Medical College Hospital
Other Study IDs: ZS-595
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Non-small Cell Lung Cancer; Leptomeningeal Metastasis
Keywords: Non-small cell lung cancer; leptomeningeal metastasis; EGFR sensitive mutations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Leptomeningeal metastasis (LM) is one of the disastrous events when managing advanced Non-small cell lung cancer (NSCLC) due to a grave prognosis. Although intrathecal (IT) chemotherapy and brain and/or spinal axis irradiation show some effects for LM in advanced NSCLC, the prognosis is still poor with median survival less than 12-14 weeks. Epidermal growth factor (EGFR) tyrosine kinase inhibitors (TKIs) showed to be effective for LM in selected NSCLC patients in some retrospective research. Our single-center prospective research indicated that the incidence of EGFR sensitive mutations (EGFRm+) in NSCLC-LM patients was high and EGFR-TKIs showed a survival benefit for LM in EGFRm+ NSCLC patients. A multi-center prospective observational biomarker study will be started in 11 lung cancer center based on our single-center prospective research result. The aims of the study are to find predictive biomarkers for LM in advanced NSCLC, to establish EGFR-TKIs based comprehensive treatment for appropriate EGFRm+ LM cases, and to establish effective clinical assessment criteria for NSCLC-LM EGFR-TKIs treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The cytological identification of malignant cells within cerebrospinal fluid (CSF).
2. Non-small cell lung cancer patients.
3. Tumor specimens or cytology specimens can be used for the EGFR gene mutation detection.
4. The entails examining cerebrospinal fluid could be obtained by lumbar puncture.
5. Expected survival time is greater than 1 month.

Exclusion Criteria:

Patients with radiologic evidence of LM not confirmed by positive CSF cytology.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Leptomeningeal metastasis (LM) in patients with non-small cell lung cancer (NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival after the diagnosis of leptomeningeal metastasis in NSCLC patients | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory Medicine, Peking Union Medical College Hospita, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xu Y, Hu M, Zhang M, Zhong W, Yin X, Sun Y, Chen M, Zhao J, Si X, Wang H, Zhang X, Zhang L, Li J, Guan H, Yang Z, Wang M. Prospective study revealed prognostic significance of responses in leptomeningeal metastasis and clinical value of cerebrospinal fluid-based liquid biopsy. Lung Cancer. 2018 Nov;125:142-149. doi: 10.1016/j.lungcan.2018.08.017. Epub 2018 Sep 17. PMID 30429013